CLINICAL TRIAL: NCT01843647
Title: Randomized, Controlled, Multicenter Study of Neoadjuvant Therapy With Icotinib in IIIA NSCLC Patients With Epidermal Growth Factor Receptor Mutation
Brief Title: Neoadjuvant Therapy of Icotinib in Epidermal Growth Factor Receptor Mutated NSCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV06
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2014-12

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Drug Therapy; Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib (Experimental): Patients receive 8-week icotinib induction treatment before surgery and 1-year icotinib adjuvant therapy after surgery.
  Interventions: Drug: Icotinib
- Chemotherapy (Active Comparator): Patients receive 8-week icotinib induction treatment before surgery and 4-cycle adjuvant chemotherapy with vinorelbine/cisplatin regimen after surgery.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Icotinib — Patients receive 8-week icotinib induction treatment before surgery and 1-year icotinib adjuvant therapy after surgery.Icotinib is administered orally with a dose 125 mg 3 times daily.
  Other Names: Commana; BPI-2009
  Arms: Icotinib
Drug: Chemotherapy — After surgery patients receive 4-cycle adjuvant chemotherapy with vinorelbine
  /cisplatin regimen, until untolerable toxicity or disease progression.
  Other Names: Vinorelbine; Cisplatin
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the overall response rate and disease free survival for IIIAN2 non-small-cell lung cancer patients with EGFR 19 or 21 exon mutation.

DETAILED DESCRIPTION:
Neoadjuvant therapy has been used for years to treat patients with non-small-cell lung cancer whose primary tumors are too large to allow for surgery. Reduction in size of the primary tumor with neoadjuvant therapy has made it possible for those patients. Moreover, the goals have expanded to include: determination of the sensitivity of the tumor so that subsequent therapy can be modified accordingly; to prolong disease free survival; to prolong survival.

ELIGIBILITY:
Inclusion Criteria:

* 1.The patients signed the written informed consent. 2.The patients present with operable IIIAN2 non-small-cell lung cancers with 19 or 21 exon mutation.

  3.The patients have no history of anti-cancer therapies including chemotherapy, radiation therapy, and surgical therapy.

  4.The patients' Eastern Cooperative Oncology Group scores are ≤ 0-1. 5.The age of patient is ≥ 18 years old with a life expectancy longer than 3 months.

Exclusion Criteria:

* 1. Patients with unresected tumor. 2. Wild EGFR type. 3. Allergic to the study drug. 4. Patients have severe non-cancerous diseases. 5. Patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 8 weeks
Disease free survival | 1 year

SECONDARY OUTCOMES:
The pathological complete response rate after neoadjuvant therapy with icotinib | 8 weeks
The lymph node staging reduction rate of patients after neoadjuvant therapy with icotinib | 8 weeks
The resection rate of patients after neoadjuvant therapy with icotinib | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China